CLINICAL TRIAL: NCT01282879
Title: Evaluation of Antifungal Prophylaxis Against Invasive Fungal Infections During Corticosteroid Containing Therapy for Graft-versus-host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Evaluation of Antifungal Prophylaxis on Graft-versus-host Disease (GVHD) Patients
Acronym: ITRAG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: In interim analysis, this study met the primary hypothesis.
Sponsor: Samsung Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: DongWhan Kim/assistant professor, Division of Hematology/Oncology, Department of Medicine,Samsung Medical Center, Sungkyunkwan University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009-08-099
Record Dates: First submitted 2011-01-23; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Graft vs Host Disease
Keywords: Itraconazole oral solution; invasive fungal infections; prophylaxis; Graft vs Host Disease; transplantation
MeSH Terms: conditions — Graft vs Host Disease; Invasive Fungal Infections | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- itraconazole, prophylaxis, Oral solution (Experimental): For GVHD patients who are required systemic glucocorticoids therapy, itraconazole oral solution will be administered at a dose of 200mg every 12 hours.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — 200mg bid, oral solution, until a dose of prednisone was tapered to 10mg/day in case of prednisone alone therapy group, or until prednisone was stopped in case of CNIs plus prednisone, CNIs plus prednisone plus mycophenolate mofetil, or mycophenolate mofetil plus prednisone group, etc.
  Other Names: Sporanox oral solution

SUMMARY:
Antifungal prophylaxis should be used in patients being treated with glucocorticoids for graft-versus-host disease (GVHD) following allogeneic hematopoietic stem-cell transplantation (HSCT). Although fluconazole has been widely used as an antifungal prophylactic agent after allogeneic HSCT, fluconazole prophlaxis only shows a limited protective role against IFIs, is not effective against invasive aspergillosis. In addition, NCCN guideline of the prevention and treatment of cancer-related infections recommends antifungal prophylaxis in patients with significant GVHD until resolution of GVHD using Posaconazole, Voriconazole, Echinocandin, or Amphotericin B. However, under the National Health Insurance System, none of the drug can be given prophylactically except itraconazole oral solution against IFIs. Itraconazole oral solution shows excellent bioavailability and good efficacy against aspergillus and fluconazole resistant candida infection.Based on these findings, we will perform prospective multicenter study evaluating the efficacy, safety and long-term outcomes of itraconazole oral solution prophylaxis against IFIs in patients treated with systemic corticosteroids for GVHD after allogeneic HSCT.

DETAILED DESCRIPTION:
Eligible patients who provided an informed consent form will be administered itraconazole oral solution (200mg bid initially, swash and swallow) in either an in patient or outpatient setting. Treatment can be initiated at the same time of or within 10 days after starting systemic immunosuppressive therapy.

Itraconazole oral solution dose can be adjusted according to the liver function test: 1) in case of - AST/ALT level 5-10 times UNL or bilirubin/ALP level 2-5 times UNL, itraconazole dose can be reduced to half (i.e. itraconazole 200mg po once daily or 100mg bid); 2) in case of - AST/ALT level > 10 times UNL or bilirubin/ALP level > 5 times UNL, itraconazole can be stopped.

GVHD treatment can be given per center's policy: With respect to acute GVHD, prednisone (1-2mg/Kg/day) oral or iv can be given on top of calcineurin inhibitor (CNI) GVHD prophylaxis. For chronic GVHD, various type of frontline regimen can be permitted including CNI+prednisone (PD), PD alone, CNI+PD+mycophenolate mofetil (MMF), or MMF+PD. Various dose of PD will be accepted if it is at least from 0.5mg/Kg/day. For example, at SMC, in case of mild grade cGVHD with high risk feature, or of moderate grade cGVHD, CNI plus PD, 0.5mg/kg/day can be given initially. In case of severe grade cGVHD, CNI plus PD, 1.0mg/Kg/day will be given.

Itraconazole will be maintained until PD is tapered to 10mg/day in case of PD alone therapy group, or until PD is stopped in case of CNI+PD or CNI+PD+MMF or MMF+PD group, etc. In addition, patients will receive itraconazole oral suspension until: 1) Development of proven or probable IFIs, 2) Severe toxicity (such as liver function abnormality - AST/ALT level > 10 times UNL or bilirubin/ALP level > 5 times UNL, 3) Worsening GVHD that requires second line therapy for steroid refractory GVHD (in this situation, investigator could stop itraconazole oral solution if there is a potential drug interaction between itraconazole oral solution and 2nd line GVHD drug or prolonged use of itraconazole oral solution could be hazardous to the patient), 4) Need to switch antifungal agent for the treatment of prolonged febrile episode related to systemic infection, thus requiring systemic antifungal treatment, 6) Withdrawal from study participation (patient's decision), or 7) Death.

ELIGIBILITY:
Inclusion Criteria:

* Patients developing or developed acute or chronic GVHD within the last 10 days which require systemic immunosuppressive therapy of corticosteroids with- or-without other immunosuppressive agents including calcineurin inhibitors.

  1. acute GVHD, grade 2-4
  2. chronic GVHD, mild grade with high risk or moderate to severe grade
* Written informed consent form

Exclusion Criteria:

* Aspartate transaminase or alanine transaminase level > 10 times UNL or Bilirubin or alkaline phosphatase level > 5 times UNL
* Active or chronic hepatitis virus B or C infection requiring antiviral therapy
* Estimated life expectancy < 30 days
* History of allergy, sensitivity, or any serious reaction to itraconazole oral solution
* Previous history of Zygomycosis
* Evidence of active fungal disease including high galactomannan titer above 0.5, within 2 weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
incidence of proven or probable invasive fungal infections | at day 100 after starting graft-versus-host disease (GVHD) treatment with corticosteroids based regimen in adjunction to itraconazole oral solution antifungal prophylaxis.

SECONDARY OUTCOMES:
safety profiles of itraconazole oral solution | during GVHD treatment with corticosteroids containing regimen
GVHD-specific survival (GSS) of patients receiving corticosteroids based GVHD treatment together with antifungal prophylaxis with itraconazole oral solution | from the onset of acute or chronic GVHD to death due to GVHD itself or GVHD-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D./Ph.D., Principal Investigator — Division of Hematology/Oncology, Department of Medicine
Locations (9):
- South Korea (9):
  - Inje University Pusan Paik Hospital, Busan, Busan
  - Gachon University Gil Hospital, Incheon, Incheon
  - Inha University Hospital, Incheon, Incheon
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Kyounggi-do
  - Samsung Medical Center, Seoul, Seoul
  - Chung-ang University Hospital, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul, Seoul

REFERENCES:
- [Background] Walsh TJ, Anaissie EJ, Denning DW, Herbrecht R, Kontoyiannis DP, Marr KA, Morrison VA, Segal BH, Steinbach WJ, Stevens DA, van Burik JA, Wingard JR, Patterson TF; Infectious Diseases Society of America. Treatment of aspergillosis: clinical practice guidelines of the Infectious Diseases Society of America. Clin Infect Dis. 2008 Feb 1;46(3):327-60. doi: 10.1086/525258. No abstract available. PMID 18177225
- [Result] Goodman JL, Winston DJ, Greenfield RA, Chandrasekar PH, Fox B, Kaizer H, Shadduck RK, Shea TC, Stiff P, Friedman DJ, et al. A controlled trial of fluconazole to prevent fungal infections in patients undergoing bone marrow transplantation. N Engl J Med. 1992 Mar 26;326(13):845-51. doi: 10.1056/NEJM199203263261301. PMID 1542320
- [Result] Winston DJ, Maziarz RT, Chandrasekar PH, Lazarus HM, Goldman M, Blumer JL, Leitz GJ, Territo MC. Intravenous and oral itraconazole versus intravenous and oral fluconazole for long-term antifungal prophylaxis in allogeneic hematopoietic stem-cell transplant recipients. A multicenter, randomized trial. Ann Intern Med. 2003 May 6;138(9):705-13. doi: 10.7326/0003-4819-138-9-200305060-00006. PMID 12729424